CLINICAL TRIAL: NCT04448405
Title: Descriptive Study on the Impact of Covid-19 Lockdown on Deviant Sexual Fantasies
Brief Title: Covid-19 Lockdown and Deviant Sexual Fantasies
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0341
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Deviant Sexual Fantasies
Keywords: sexuality; Confinement; sex offender; outcome; paraphilia; cybersexuality
MeSH Terms: conditions — Sexuality; Paraphilic Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients followed by the CRIAVS: Patients followed by the CRIAVS (resource center for workers working with authors of sexual violence) in CHU Motpellier from June to October 2020
  Interventions: Behavioral: Questionnaire for evaluation of confinement on deviant sexual fantasies

INTERVENTIONS:
Behavioral: Questionnaire for evaluation of confinement on deviant sexual fantasies — Questionnaire for evaluation of confinement on deviant sexual fantasies. Population already followed for deviant fantasies

SUMMARY:
Our society is going through an unprecedented situation: the COVID 19 Pandemic is forcing many populations, worldwide, into confinement for their own protection. The very characteristics of this confinement and of the disease (isolation, potential severity of the illness, being psychologically unprepared for such a circumstance) have a significant impact on one's psyche, like emotional disorders -anxiety/depression-, difficulties when returning to normal life, vicarious traumas… Confinement is paradoxical in as although well-intended to protect the individual, it leads to the isolation of the individual. This paradox is destabilizing one's feelings, because when the investigators feel the need for protection and reassurance, the investigators are left alone and feel abandoned. The investigators therefore understand that this confinement framework is in essence a situation that might revive unresolved deprivation situations from the childhood. How to react in front of this upsurge in anxiety? Strategies used may include, among others, escape in the imaginary through numerical tools or others, and /or going to the actual characterized by deviant sexual behaviours. The investigators know in fact that certain moments, like anxiety, depression, boredom, psychological unrest are propicious for acting, for violent sexual offenders. The investigators therefore pay extra attention to our patients in such periods favoring these kinds of trouble.

This study will enable us to understand if the confinement associated with COVID 19 has generated anxiety that lead sexual offenders or individuals with paraphilic disorders to engage into deviant fantasies or, potentially sexual activities.

DETAILED DESCRIPTION:
The questionnaire is handed only one time to each patient and the questions it contains are part of those commonly used.

How do the investigators precisely operate: self questionnaire on paper, handed to each patient followed by the CRIAVS in the waiting room, and returned by the patient to the therapist, or the department, in a sealed envelope. Digital data collection thereafter.

ELIGIBILITY:
Inclusion criteria:

* Adults
* Consulting at the CRIAVS between June and end October 2020

Exclusion criteria:

* no demance
* no decompensated psychatric disorder
* no tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed by the CRIAVS (resource center for workers working with authors of sexual violence) in CHU Motpellier from June to October 2020
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Impact of confinement on deviant fantasies | through study completion, an average of 1 year
  Lickert scale from 1 to 10

SECONDARY OUTCOMES:
Intensity of deviant fantasies | through study completion, an average of 1 year
  Likert scale from 0 to 10
Frequency of deviant fantasies | through study completion, an average of 1 year
  Likert scale from 0 to 10
Paraphilic type impacted | through study completion, an average of 1 year
  Box to be chacked by the patient: exhibition, voyeurism, pedophilia, sadomasochism, crossdressing, raptophilia
Occurrence of sexual act | through study completion, an average of 1 year
  Number given by the patient
Access mode for deviant fantasies | through study completion, an average of 1 year
  Did you use internet : yes or no
Use of support during confinement | through study completion, an average of 1 year
  box yes or no Was support different? Did you use remote consultation? How did you like it?
Evaluating anxiety/depression level | through study completion, an average of 1 year
  HAD Hospital Anxiety And Depression Scale The HAD scale is an instrument for detecting anxiety and depressive disorders. It has 14 listed items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), two scores are obtained (maximum score for each score = 21). - 7 or less: absence of symptoms
  - 8 to 10: doubtful symptomatology - 11 and more: certain symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Celine BAIS, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC